CLINICAL TRIAL: NCT05810857
Title: Comparative Effects of Motor Relearning Programme Versus Mirror Therapy on Balance and Gait in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/525
Record Dates: First submitted 2023-03-18; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Relearning Program (Other)
  Interventions: Diagnostic Test: Motor Relearning Program
- Mirror Therapy (Other)
  Interventions: Diagnostic Test: Mirror Therapy

INTERVENTIONS:
Diagnostic Test: Motor Relearning Program — patients will receive Motor Relearning Program including static and dynamic sitting and standing balance while static sitting balance
  Arms: Motor Relearning Program
Diagnostic Test: Mirror Therapy — "Mirror Therapy" protocol. The baseline treatment will be weight bearing in standing which is extension of knee and weight bearing in standing on inclined
  Arms: Mirror Therapy

SUMMARY:
To determine the effect of Motor Relearning Program versus Mirror Therapy for balance and gait in chronic ischemic stroke patients

ELIGIBILITY:
Inclusion Criteria:

* • Chronic ischemic stroke of six or more than six months.

  * Patients with age - 45- 65 years.
  * Patients with good cognitive status i.e. 20 or more on MMSE.(Mini Mental Status Examination).
  * Patients of both genders
  * Patients with ambulation before stroke.

Exclusion Criteria:

* • Patients who have musculoskeletal disorder impending lower limb function.

  * Patient with any other Neurological disease.
  * Patients have severe lower limb deformities, and vestibular disorders.
  * Patients who have any joint disorder of lower limb.
  * Patients who have any cardiac problem.
  * Patients with history of recurrent stroke.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Mirror Therapy Techinique, Motor Relearning Programme Techinique | 6 Months

IPD SHARING:
Plan to Share IPD: No